CLINICAL TRIAL: NCT02631850
Title: Video Game Rehabilitation for Outpatient Stroke (VIGoROUS): A Multi-center Comparative Effectiveness Trial of In-home Gamified Constraint-induced Movement Therapy for Rehabilitation of Chronic Upper Extremity Hemiparesis.
Brief Title: Effectiveness of Virtual Reality Gaming Therapy Versus CI Therapy for Upper Extremity Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: OhioHealth (Other); Providence Medical Research Center (Other); University of Alabama at Birmingham (Other); University of Massachusetts, Lowell (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Deborah S Larsen, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012H0151
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Hemiparesis
Keywords: Constraint-induced movement therapy; gaming; virtual reality; upper extremity; CI therapy; rehabilitation; stroke; hemiparesis; therapy; self-management; in-home; remote; telerehabilitation
MeSH Terms: conditions — Stroke; Paresis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Traditional CI Therapy (Active Comparator): Participants will receive a 35-hour "dose" of CI therapy. Treatment will consist of 35 therapist/client contact hours in the clinic, 10 weekdays, over 3 weeks. To promote carry-over of motor gains to daily activities, participants will complete: (1) a treatment contract, (2) daily self-report of arm use, and (3) problem-solving to overcome barriers to use of the more affected upper extremity. In addition, the client will agree to wear a padded restraint mitt on the less affected hand for the majority of waking hours to encourage use of the weaker hand for daily activities. Finally, the participant will agree to 30 minutes per day of individualized task-practice outside the clinic (in addition to training in the clinic) focused on functional activities catered towards accomplishing the person's therapeutic goals.
  Interventions: Behavioral: Traditional CI Therapy
- Gaming CI Therapy (Active Comparator): 15 hours of progressive massed motor practice will occur through in-home video game play over 15 consecutive weekdays. Participants will play the game during times of their choosing. The participant will wear an activity monitor biofeedback device for the majority of waking hours. As with traditional CI therapy, the client will agree to an additional 30 minutes per day of individualized task-practice. Five therapist/client contact hours will occur in the clinic on approximate treatment days 1, 3, 6, and 11 and will focus on treatment elements that cannot be readily addressed through the game, such as problem-solving to help the participant carry over motor gains to daily life.
  Interventions: Behavioral: Gaming CI Therapy
- Gaming CI Therapy with Additional Contact via Video Conference (Active Comparator): This group will receive treatment that is identical to Group 2, but will receive an additional 2.6 hours video conference consultation throughout the treatment period.
  Interventions: Behavioral: Gaming CI Therapy with Additional Contact via Video Conference
- Traditional Occupational Therapy/Physical Therapy (Active Comparator): Five therapist/client contact hours will occur on approximate treatment days 1, 3, 6, and 11 (same schedule as gaming CI therapy). 1 hour progressive resistance exercise to establish and progress an upper extremity home exercise program, 2 hours of neuromuscular reeducation, and 2 hours functional practice on activities of daily living (ADLs) with verbal encouragement to use the more affected upper extremity to the largest extent possible. Home practice consists of strengthening exercises, designed to increase range of motion, prescribed twice daily. After completing their participation in the standard OT condition (6 months), participants will be crossed-over to a CI therapy gaming only condition. This condition will be identical to that described above, excluding therapist contact throughout the intervention. Rather, participants will receive a DVD explaining the intervention and guiding them through use of the system.
  Interventions: Behavioral: Traditional Occupational Therapy/Physical Therapy

INTERVENTIONS:
Behavioral: Traditional CI Therapy — Intensive in-person therapy for upper extremity hemiparesis.
  Arms: Traditional CI Therapy
Behavioral: Gaming CI Therapy — Intensive remote (via video game) therapy for upper extremity hemiparesis.
  Arms: Gaming CI Therapy
Behavioral: Gaming CI Therapy with Additional Contact via Video Conference — Intensive remote (via video game) therapy for upper extremity hemiparesis with additional therapist contact via video conference.
  Arms: Gaming CI Therapy with Additional Contact via Video Conference
Behavioral: Traditional Occupational Therapy/Physical Therapy — Traditional in-person therapy focusing on the rehabilitation of the upper extremity.
  Arms: Traditional Occupational Therapy/Physical Therapy

SUMMARY:
The current proposal aims to conduct a multi-site randomized controlled trial comparing virtual-reality gaming delivery of Constraint Induced Movement therapy (CI therapy) with (1) traditional clinic-based CI therapy of equal total active therapy duration and (2) a control group equating the dose of in-person therapy. Individuals with chronic stroke will be randomized to one of four different interventions: (1) traditional clinic-based CI therapy (35 therapist/client contact hours), (2) therapist-as-consultant virtual reality CI therapy (5 therapist/client contact hours in the clinic and 15 hours of independent game play at home), (3) therapist-as-consultant virtual reality CI therapy with additional therapist contact via telerehabilitation (5 therapist/client contact hours in the clinic, 2.6 therapist contact hours via teleconference, and 15 hours of independent game play in the home), and (4) 5 hours of standard occupational therapy (OT) / physical therapy (PT). After 6-month follow-up, individuals assigned to standard OT/PT will cross over to a modified gaming therapy condition (a stand-alone application of the rehabilitation game without additional therapist contact).

DETAILED DESCRIPTION:
Detailed study description published in BMC Neurology (2017).

ELIGIBILITY:
Inclusion Criteria:

* Males, females, or any gender identity 18 years of age or older
* Experienced a stroke resulting in mild-to-moderate hemiparesis at least six months prior to enrollment (suggested range of motion (ROM) criteria includes: 45° shoulder abduction and flexion, 20° elbow extension, 20° wrist extension, and 10° extension of thumb and finger)
* Have preserved ability to comprehend and participate in basic elements of the therapy

Exclusion Criteria:

* Concurrent participation in other experimental trials for motor dysfunction treatment
* Receiving Botox therapy currently or in the past 3 months
* Have medical conditions that would place volunteers at higher risk of adverse events (e.g., renal disease, frailty, pregnancy, dementia, severe pain, end-stage/degenerative diseases)
* Have received intensive upper-extremity rehabilitation in the chronic phase post-stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Larsen, PhD, Principal Investigator — The Ohio State U.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Missouri, Columbia, Missouri
  - The Ohio State University, 2154 Dodd Hall, Columbus, Ohio
  - OhioHealth Rehabilitation, Columbus, Ohio
  - Providence Medford Medical Center, Medford, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Data will be made public upon publication.
Supporting Information: Study Protocol, ICF
Time Frame: Upon publication of the main results paper.
Access Criteria: Will update with public URL upon acceptance of the study paper. Prior to this, those interesting in accessing the study data can contact lynne_gauthier@uml.edu to arrange access.

REFERENCES:
- [Background] Gauthier LV, Kane C, Borstad A, Strahl N, Uswatte G, Taub E, Morris D, Hall A, Arakelian M, Mark V. Video Game Rehabilitation for Outpatient Stroke (VIGoROUS): protocol for a multi-center comparative effectiveness trial of in-home gamified constraint-induced movement therapy for rehabilitation of chronic upper extremity hemiparesis. BMC Neurol. 2017 Jun 8;17(1):109. doi: 10.1186/s12883-017-0888-0. PMID 28595611
- [Derived] Gauthier LV, Ravi R, DeLuca D, Zhou W. Dose Response to Upper Extremity Stroke Rehabilitation Varies by Individual: Early Indicators of Treatment Response. Stroke. 2024 Mar;55(3):696-704. doi: 10.1161/STROKEAHA.123.045039. Epub 2024 Feb 26. PMID 38406850
- [Derived] Borstad A, Nichols-Larsen D, Uswatte G, Strahl N, Simeo M, Proffitt R, Gauthier L. Tactile Sensation Improves Following Motor Rehabilitation for Chronic Stroke: The VIGoROUS Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Aug;36(8):525-534. doi: 10.1177/15459683221107893. Epub 2022 Jun 11. PMID 35695197
- [Derived] Gauthier LV, Nichols-Larsen DS, Uswatte G, Strahl N, Simeo M, Proffitt R, Kelly K, Crawfis R, Taub E, Morris D, Lowes LP, Mark V, Borstad A. Video game rehabilitation for outpatient stroke (VIGoROUS): A multi-site randomized controlled trial of in-home, self-managed, upper-extremity therapy. EClinicalMedicine. 2021 Dec 17;43:101239. doi: 10.1016/j.eclinm.2021.101239. eCollection 2022 Jan. PMID 34977516
- [Derived] Rafiei MH, Kelly KM, Borstad AL, Adeli H, Gauthier LV. Predicting Improved Daily Use of the More Affected Arm Poststroke Following Constraint-Induced Movement Therapy. Phys Ther. 2019 Dec 16;99(12):1667-1678. doi: 10.1093/ptj/pzz121. PMID 31504952

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 193 participants met enrollment criteria and signed a consent form during the screening visit. 14 withdrew shortly thereafter, citing logistical challenges (e.g., scheduling, transportation). 5 no-showed to the first treatment session and could not be reached. 4 experienced medical events that prompted them to withdraw prior to beginning treatment. 2 could not be contacted to schedule participation. The randomization assignment was recycled back into pool for those who did not begin treatment.
Groups:
- Traditional Occupational Therapy/Physical Therapy: Five therapist/client contact hours will occur on approximate treatment days 1, 3, 6, and 11 (same schedule as gaming CI therapy). 1 hour progressive resistance exercise to establish and progress an upper extremity home exercise program, 2 hours of neuromuscular reeducation, and 2 hours functional practice on ADLs with verbal encouragement to use the more affected upper extremity to the largest extent possible. Home practice consists of strengthening exercises, designed to increase range of motion, prescribed twice daily. After completing their participation in the standard OT condition (6 months), participants will be crossed-over to a CI therapy gaming only condition. This condition will be identical to that described above, excluding therapist contact throughout the intervention. Rather, participants will receive a DVD explaining the intervention and guiding them through use of the system.
  Traditional Occupational Therapy/Physical Therapy: Traditional in-person therapy focusing on the rehabilitation of the upper extremity.
Period: Treatment Period
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Started | 41 (One participant was withdrawn during treatment because medical records review revealed that the motor deficit was due to an old orthopedic injury and not stroke. This participant had experienced a Transient Ischemic Attack, but no stroke that resulted in lasting neurological motor deficit. 40 participants were thus analyzed for this group in the intent-to-treat analysis even though 41 began treatment.) | 44 | 45 | 38
Completed | 38 | 38 | 41 | 33
Not Completed | 3 | 6 | 4 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 2 | 3
Not completed — Family medical issue | 1 | 0 | 0 | 0
Period: 6 Month Follow up
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Started | 38 | 38 | 41 | 33
Completed | 31 | 25 | 35 | 22
Not Completed | 7 | 13 | 6 | 11
Not completed — Lost to Follow-up | 5 | 8 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 4 | 1 | 3
Not completed — moved out of state, transportation issues, family medical issue | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Includes all eligible participants that began treatment.
Groups:
- Gaming CI Therapy With Additional Contact Via Video Conference: This group will receive treatment that is identical to Group 2, but will receive an additional 4 hours video conference consultation throughout the treatment period.
  Gaming CI Therapy with Additional Contact via Video Conference: Intensive remote (via video game) therapy for upper extremity hemiparesis with additional therapist contact via video conference.
- Traditional Occupational Therapy/Physical Therapy: Five therapist/client contact hours will occur on approximate treatment days 1, 3, 6, and 11 (same schedule as gaming CI therapy). 1 hour progressive resistance exercise to establish and progress an upper extremity home exercise program, 2 hours of neuromuscular reeducation, and 2 hours functional practice on ADLs with verbal encouragement to use the more affected upper extremity to the largest extent possible. Home practice consists of stretching exercises, designed to increase range of motion, prescribed twice daily. After completing their participation in the standard OT condition (6 months), participants will be crossed-over to a CI therapy gaming only condition. This condition will be identical to that described above, excluding therapist contact throughout the intervention. Rather, participants will receive a DVD explaining the intervention and guiding them through use of the system.
  Traditional Occupational Therapy/Physical Therapy: Traditional in-person therapy focusing on the rehabilitation of the upper extremity.
- Total: Total of all reporting groups
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy | Total
Number analyzed (Participants) | 40 | 44 | 45 | 38 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13) | 60 (14) | 56 (17) | 63 (14) | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 19 | 8 | 57
  Male | 30 | 24 | 26 | 30 | 110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 14 | 9 | 10 | 42
  White | 29 | 27 | 30 | 24 | 110
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 2 | 8
Time since stroke [Mean (Standard Deviation); unit: years] — Chronicity calculated by subtracting the date of stroke from the date of pre-test.
  years | 4.9 (9.8) | 5.2 (6.5) | 3.4 (5.1) | 5.8 (8.1) | 4.8 (7.6)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The MoCA is a cognitive screening tool. Scores on this measure range from 0-30 and reflect the number of items successfully answered; +1 point is given for <12 years of education. Items assess language, executive function, memory, orientation, and visuoconstruction ability. Below 24 indicates mild cognitive impairment. Below 16 indicates more severe cognitive impairment (e.g., may indicate dementia).
  units on a scale | 21.6 (6.4) | 22.3 (5.4) | 22.5 (5.6) | 20.1 (6.0) | 21.7 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test
Description: Assesses the time to complete 15 standardized tasks (e.g., folding a towel, stacking checkers, placing hand on top of a box). Items that cannot be accomplished score 120 seconds. Times are natural log transformed to reflect proportional improvement (approximate % change) and correct for skew. On the log transformed scale, -.22 reflects normal ability, 4.79 = can't accomplish task. For improvement in mean log transformed performance time, -4.79 = best possible improvement, 0 = no improvement, positive scores = worsening. A proportional improvement of 16% (mean log transformed performance time change = -.17) is considered clinically meaningful.
Time Frame: 0 to 1 months
Population: Modified intent-to-treat (those who started treatment)
Measure: Mean (Standard Deviation); unit: natural log of performance time change
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 41 | 44 | 45 | 38
natural log of performance time change | -0.38 (0.35) | -0.24 (0.33) | -0.29 (0.33) | -0.22 (0.36)

2. Primary Outcome: Motor Activity Log Quality of Movement Scale
Description: Assessment evaluates the amount and quality of everyday arm use. The scale consists of 28 activities of daily living (e.g., washing hands, drinking from a cup). Participants self-report on an 11-point scale (0-5 with half-point increments, 0=not attempted to 5=attempted with normal movement). The total score on the measure reflects the mean of the individual item scores. A change of 1.0 on the scale is considered clinically meaningful.
Time Frame: 0 to 1 months
Population: Modified intent-to-treat (those who started treatment)
Measure: Mean (Standard Deviation); unit: change in mean MAL
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 40 | 44 | 45 | 38
change in mean MAL | 1.7 (.7) | 1.3 (.7) | 1.5 (.7) | .5 (.6)

3. Secondary Outcome: Change in Neuro-Quality of Life (Neuro-QOL)
Description: Computerized adaptive assessment on several domains of quality of life: sleep, mobility, positive affect and well-being, fatigue, satisfaction with social roles, cognitive function, anxiety, and communication. Neuro-QOL uses a T score which has a mean of 50 and SD of 10, based on the norming sample used. All Neuro-QOL banks and scales are scored such that a higher score reflects more of what is being measured. Scores are reported as mean T-scores across the assessed domains. Positive changes indicate an improvement.
Time Frame: 0 to 1 months
Population: Modified intent-to-treat
Measure: Mean (Standard Deviation); unit: Mean change in T-score
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 40 | 44 | 45 | 38
Mean change in T-score | .69 (2.13) | -.05 (1.66) | -.72 (2.49) | .82 (2.95)

4. Secondary Outcome: Bilateral Activity Monitors
Description: Devices to monitor upper extremity movement are worn throughout treatment. The devices count movements made with each arm, defined as an acceleration of 2g for at least 500 ms. The ratio of more affected to less affected arm use is then calculated for each treatment day. The best linear fit trajectory for each participant is calculated after removal of outliers. The treatment change reported here reflects the difference between the best-fit-line at post-treatment and the best-fit-line at pre-treatment. Positive change indicates improvement.
Time Frame: 0 to 1 month
Population: Those for whom accelerometer data was obtained bilaterally.
Measure: Mean (Standard Deviation); unit: change in ratio of arm use
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 15 | 21 | 22 | 19
change in ratio of arm use | .12 (.21) | 0 (.25) | .05 (.20) | .04 (.30)

5. Secondary Outcome: Change in Brief Kinesthesia Test (BKT)
Description: This measures was intended to measure proprioception in the upper extremity; however, performance on the measure is also known to be adversely affected by motor impairment. The experimenter guides individuals along movement trajectories between 2 and 9 inches with their vision obscured. They are then asked to reproduce the movement trajectories. The summed difference between the desired and produced trajectory endpoints in cm is reported. A negative change indicates an improvement.
Time Frame: 0 to 1 months
Measure: Mean (Standard Deviation); unit: sum of vector distances in cm
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 40 | 44 | 45 | 38
sum of vector distances in cm | -1.8 (6.6) | -.9 (4.2) | .8 (4.6) | -1.0 (6.3)

6. Secondary Outcome: Semmes-Weinstein Monofilament Test
Description: Sensory evaluator of touch sensation. Units are the log transformed grams of pressure detected by the index finger of the paretic hand. Scores range from -1.8 to 5.7. Smaller scores indicate better sensation. Negative change indicates improvement.
Time Frame: 0 to 1 months
Population: Modified intent-to-treat
Measure: Mean (Standard Deviation); unit: change in log grams
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 40 | 44 | 45 | 38
change in log grams | -.25 (1.11) | -.39 (1.66) | -.03 (1.90) | -.50 (1.93)

7. Secondary Outcome: 9 Hole Peg Test
Description: Assessment to measure upper extremity distal motor function. The assessment measures the time to place 9 pegs into grooves on a board. Due to the inability of a majority of the participants to place all 9 pegs during the 120 seconds allotted for the test, performance was transformed into a rate metric to reduce floor effects. The outcome is expressed as change in the number of pegs per minute.
Time Frame: 0 to 1 months
Population: Modified intent-to-treat
Measure: Mean (Standard Deviation); unit: change in pegs per minute
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 40 | 44 | 45 | 38
change in pegs per minute | -.08 (3.36) | -.53 (3.27) | .49 (2.61) | .94 (4.40)

8. Other Pre Specified Outcome: Montreal Cognitive Assessment (MoCA)
Description: Assessment to measure cognitive function at baseline. The range of the MoCA assessment is 0-30. Scores below 24 indicate cognitive impairment and scores below 16 indicate severe cognitive impairment. The MoCA was administered for the purpose of characterizing the study population and was examined as a potential covariate in linear mixed effect models examining primary and secondary outcome measures.
Time Frame: baseline only measure, exploratory covariate in the analysis
Population: Those who started treatment
Measure: Mean (Standard Deviation); unit: Total score at baseline
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
Number analyzed (Participants) | 40 | 44 | 45 | 38
Total score at baseline | 21.6 (6.4) | 22.3 (5.4) | 22.5 (5.6) | 20.1 (6.0)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Traditional CI Therapy | Gaming CI Therapy | Gaming CI Therapy With Additional Contact Via Video Conference | Traditional Occupational Therapy/Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/45 | 0/44 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/45 | 0/44 | 0/38
Other Adverse Events (participants affected / at risk) | 0/41 | 1/45 | 0/44 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional CI Therapy (N=41) | Gaming CI Therapy (N=45) | Gaming CI Therapy With Additional Contact Via Video Conference (N=44) | Traditional Occupational Therapy/Physical Therapy (N=38)
bruising on wrist from wearing monitoring watch too tight (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT02631850/Prot_SAP_ICF_000.pdf